CLINICAL TRIAL: NCT05133518
Title: A Phase 2, Factorial-Designed, Randomized, Double-Blind, Placebo-Controlled, Parallel- Cohort Study to Evaluate Efficacy and Safety of MELT-300 and the Contribution of Midazolam and Ketamine Components to Sedation and Intraoperative Ocular Analgesia in Subjects Undergoing Cataract Extraction With Lens Replacement (CELR)
Brief Title: A Study of MELT-300 (Midazolam and Ketamine Sublingual Tablets) for Sedation and Intraoperative Ocular Analgesia in Participants Undergoing Cataract Extraction With Lens Replacement (CELR)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Melt Pharmaceuticals (Industry)
Collaborators: Worldwide Clinical Trials (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MELT-2-001
Record Dates: First submitted 2021-11-12; First posted 2021-11-24 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Cataract
Keywords: Cataract surgery; Intraocular pressure; Intraoperative ocular pain; Sedation; Lens replacement; MELT-300; Cataract extraction
MeSH Terms: conditions — Cataract | interventions — Midazolam; Ketamine

STUDY DESIGN:
Intervention Model Description: Factorial-designed, randomized, double-blind, placebo-controlled, parallel-cohort safety and efficacy study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MELT-300 (Active Comparator): Participants will receive a single dose of MELT-300 sublingual, rapidly dissolving tablet containing 3 mg of midazolam and 50 mg of ketamine.
  Interventions: Drug: MELT-300
- Midazolam alone (Active Comparator): Participants will receive a single dose of midazolam 3 mg sublingual tablet.
  Interventions: Drug: Midazolam alone
- Ketamine alone (Active Comparator): Participants will receive a single dose of ketamine 50 mg sublingual tablet.
  Interventions: Drug: Ketamine alone
- Placebo (Placebo Comparator): Participants will receive a single dose of a matching placebo sublingual tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MELT-300 — Sublingual tablet
  Arms: MELT-300
Drug: Midazolam alone — Sublingual tablet
  Arms: Midazolam alone
Drug: Ketamine alone — Sublingual tablet
  Arms: Ketamine alone
Drug: Placebo — Sublingual tablet
  Arms: Placebo

SUMMARY:
The primary purpose of the study is to evaluate the efficacy and safety of MELT-300 (Midazolam and Ketamine Sublingual Tablets) and the contribution of midazolam and ketamine components to sedation and during the surgery or ocular analgesia in participants undergoing cataract surgery with lens replacement.

DETAILED DESCRIPTION:
This is a Phase 2, factorial-designed, randomized, double-blind, placebo-controlled, parallel-cohort study to be conducted in 324 adult male and female participants who are ≥ 55 years of age and undergoing cataract extraction with lens replacement. An additional 3 participants per site (first 3 participants enrolled per site) will be considered sentinel participants for the purpose of ensuring safety and that logistical and operational challenges that may occur during the study are identified and mitigated. Sentinel participants will be evaluated for safety but not for efficacy. The study aims to evaluate the efficacy and safety of MELT-300 and the contribution of midazolam and ketamine components for procedural sedation prior to cataract surgery. In the study, eligible study participants will be randomly assigned (1:1:1:1 ratio) to one of the following treatments: MELT-300 (3 mg/50 mg), midazolam 3 mg, ketamine 50 mg, and placebo sublingual tablet 30 (± 5) minutes prior to the anticipated start of surgery (defined as instillation of topical ocular anesthetic drops [i.e., proparacaine]) without food or water in the operating room. At the time of dosing, participants will be instructed to hold the tablet under their tongue until it is completely dissolved and to not swallow or chew the tablets. The study duration will be up to 35 days, including 28 days for screening and 7 ± 2 days after surgery.

Efficacy assessments will be performed after study medication administration before surgery, intraoperatively, and postoperatively on Day 1 (end of surgery defined as drape removal). Efficacy assessments will include assessments of sedation and intraoperative pain, the need for rescue medication for sedation or pain, and the ability to complete the surgery. Safety will be monitored at baseline, intraoperatively, postoperatively on Day 1, on the day after surgery (Day 2, via a phone call), and at 1 week (Day 8 ± 2 days) after dosing of study medication. Safety assessments will include monitoring of AEs, vital sign measurements, physical examinations, and 12-lead ECGs. Exploratory endpoints are postoperative pain as measured by the NPRS prior to discharge, 6 hours +/- 30 minutes after the end of surgery on Day 1 and on Days 2 (the day after surgery), the percentage of participants with concomitant medication opioid use, and average opioid consumption on Day 2 and participant likelihood of wanting study drug again for second cataract surgery as measured by an 11-point Likert scale on Day 2.

ELIGIBILITY:
Inclusion Criteria:

1. Are to undergo unilateral primary uncomplicated CELR under topical anesthesia, with a phacoemulsification device and insertion of an intraocular lens.

Exclusion Criteria:

1. Participants scheduled for simultaneous bilateral or 2nd-eye cataract surgery (note, subjects scheduled for a future 2nd eye cataract study are eligible for the study).
2. Known sensitivity to benzodiazepines or ketamine.
3. Known sensitivity to -caines (including proparacaine), benzalkonium chloride (BAK).
4. Intraocular pressure (IOP) ≥ 23 mmHg in the study eye and/or ≥ 30 mmHg in the fellow eye at screening. This IOP exclusion requirement will only need to be re-confirmed on the day of surgery if it has been > 14 days since the screening visit.
5. History of iritis, or any ocular trauma with iris damage in the study eye.
6. Presence of active corneal pathology other than corneal pathology per slit lamp and an external eye exam at screening in either eye.
7. Presence of extraocular/intraocular inflammation in either eye.
8. Presence of active bacterial and/or viral infection in either eye.
9. History of intraocular non-laser surgery in the study eye within the 3 months prior to day of surgery, or intraocular laser surgery in the study eye within 30 days prior to the day of surgery.
10. Require or are planning other additional ocular surgery during the cataract surgery.

12. Have a history or clinical manifestations (e.g., signs, symptoms, laboratory values, diagnostic imaging, etc.) of significant gastrointestinal, cardiovascular, hepatic, renal, hematological, endocrine, neurological, psychiatric, respiratory, or other medical condition that in the opinion of the investigator might confound the study results or pose additional risk in administering the study procedures.

13. History of or presence of any connective tissue disorder (i.e., lupus, rheumatoid arthritis, fibromyalgia).

14. Use of disallowed medications, including the following:

1. Pain medication (opioids, non-steroidal anti-inflammatory drugs [NSAIDs], cyclooxygenase-2 [COX-2] inhibitors, tramadol, ketamine, clonidine, gabapentin, pregabalin, or cannabinoids) within 3 days prior to Day 1, or routine, daily opioid therapy within the past 30 days.
2. Central nervous system (CNS) active drugs such as benzodiazepines, tricyclic antidepressants, serotonin, and norepinephrine reuptake inhibitors (SNRIs), or selective serotonin reuptake inhibitors (SSRIs) for pain within 7 days prior to Day 1. These drugs are permitted for non-pain indications if the dose has been stable for at least 30 days prior to Day 1 and is planned to remain stable throughout the study. The use of lorazepam and other sleep medications, except those containing analgesic properties, is permitted.
3. Use of parenteral or oral corticosteroid(s) within 14 days prior to Day 1.
4. Antihypertensive agent or diabetic regimen at a dose that has not been stable for at least 30 days, or which is not expected to remain stable throughout the study.

   15. Chronic pain rated moderate to severe within the past week (4-pt categorical scale, 0=no pain, 1=mild pain, 2=moderate pain, 3=severe pain). 17. Hospital Depression and Anxiety Scale (HADS) score > 10

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-11-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Success for Procedural Sedation by Using Ramsay Sedation Scale | Day 1
  The Ramsay Sedation Scale (RSS) was the first scale to be defined for the sedated participants and was designed as a test of arousability. The Ramsay Scale provides three levels of 'awake' states (score 1-3) and three levels of 'asleep' states (score 4-6). A score of 2 (participant is cooperative, orientated, and tranquil) best fits an optimum sedation level based on the criteria of calm, comfortable, communicative, and cooperative participants.
  Ramsay Sedation Scale
  1. =Participant is anxious and agitated or restless, or both
  2. =Participant is cooperative, oriented, and tranquil
  3. =Participant responds to commands only
  4. =Participant exhibits brisk response to a light glabellar tap or loud auditory stimulus
  5. =Participant exhibits a sluggish response to a light glabellar tap or loud auditory stimulus
  6. =Participants exhibits no response RSS score will be assessed pre-operatively, intra-operatively, and post-operatively on Day 1
Mean Intraoperative Analgesia as Measured by the Numeric Pain Rating Scale | Intraoperatively on Day 1
  The Numeric Pain Rating Scale (NPRS) is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")

SECONDARY OUTCOMES:
Percentage of Pre-operative Target Sedation Responders by Ramsay Sedation Scale (level 2 or 3) | Pre-operatively (at baseline), intra-operatively and post-operatively on Day 1
  The Ramsay Sedation Scale (RSS) was the first scale to be defined for the sedated participants and was designed as a test of arousability. The Ramsay Scale provides three levels of 'awake' states (score 1-3) and three levels of 'asleep' states (score 4-6). A score of 2 (participant is cooperative, orientated, and tranquil) best fits an optimum sedation level based on the criteria of calm, comfortable, communicative, and cooperative participants.
  Ramsay Sedation Scale
  1. =Participant is anxious and agitated or restless, or both
  2. =Participant is cooperative, oriented, and tranquil
  3. =Participant responds to commands only
  4. =Participant exhibits brisk response to a light glabellar tap or loud auditory stimulus
  5. =Participant exhibits a sluggish response to a light glabellar tap or loud auditory stimulus
  6. =Participants exhibits no response
Percentage of Analgesia Responders Using Numeric Pain Rating Scale | Pre-operatively (at baseline), intra-operatively and post-operatively on Day 1
  The Numeric Pain Rating Scale (NPRS) is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Number of Participants with Sedation Scores | After study medication administration before surgery (baseline), intraoperatively, and postoperatively on Day 1 (end of surgery defined as drape removal)
  The Ramsay Sedation Scale (RSS) was the first scale to be defined for the sedated participants and was designed as a test of arousability. The Ramsay Scale provides three levels of 'awake' states (score 1-3) and three levels of 'asleep' states (score 4-6). A score of 2 (participant is cooperative, orientated, and tranquil) best fits an optimum sedation level based on the criteria of calm, comfortable, communicative, and cooperative participants.
  Ramsay Sedation Scale
  1. =Participant is anxious and agitated or restless, or both
  2. =Participant is cooperative, oriented, and tranquil
  3. =Participant responds to commands only
  4. =Participant exhibits brisk response to a light glabellar tap or loud auditory stimulus
  5. =Participant exhibits a sluggish response to a light glabellar tap or loud auditory stimulus
  6. =Participants exhibits no response
Number of Participants with Pain Scores | Before dosing on the day of surgery (Day 1)
Number of Participants-rated Worst Pain Following Completion of Surgery | Pre-operatively (at baseline), intra-operatively, and post-operatively on Day 1
Percentage of Participants Able to Complete Surgery | Pre-operatively (at baseline), intra-operatively and post-operatively on Day 1
Percentage of Participants Without Interruption of Surgery for Intervention (Other Than Rescue Medication) Due to Pain or Anxiety | Pre-operatively (at baseline), intra-operatively, and post-operatively on Day 1
Percentage of Participants Requiring Rescue Sedative Medication | Pre-operatively (at baseline) and Intra-operatively on Day 1
  The preoperative target level of sedation for this trial is Ramsay Sedation Scale (RSS) 2 or 3. If a participant does not achieve this level of sedation prior to the start of surgery (administration of topical local anesthesia), rescue sedation medication (i.e., intravenous midazolam only, at a dose determined by Investigator or anesthesiologist) may be given. Use of rescue sedation medication during surgery will be allowed if a participant's RSS score is <2.
Percentage of Participants Requiring Rescue Analgesic Medication | After study medication administration before surgery (baseline) and intraoperatively
  Intraoperative pain assessments using the Numeric Pain Rating Scale (NPRS) scale, from 0 (no pain) to 10 (extreme pain), will be assessed.
  The NPRS is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Number of Participants Reported with At least One Treatment Emergent Adverse Event (TEAE) | Pre-operatively (at baseline), intra-operatively post-operatively on Day 1, on the day after surgery (Day 2, via a phone call), and at 1 week (Day 8 ± 2 days) after dose of study medication
  A treatment-emergent adverse event is defined as any event not present prior to the initiation of the drug treatment or any event already present that worsens in either intensity or frequency following exposure to the drug treatment.

OTHER OUTCOMES:
Postoperative Pain as measured by the Numeric Pain Rating Scale Scores | Prior to discharge, 6 hours +/- 30 minutes, and on Day 2 (the day after surgery)
  The Numeric Pain Rating Scale (NPRS) is a segmented numeric version of the Visual Analog Scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain. The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable").
Percentage of Participants with Concomitant Medication Opioid Use and Average Opioid Consumption | Day 2
  Concomitant medication is a medication, a person is taking that is not being studied in the clinical trial he or she is taking part in.
Participant Likelihood of Wanting Study Drug Again for Second Cataract Surgery as Measured by 11-point Likert Scale | Day 2
  A Likert Scale is a Psychometric Scale commonly involved in research that employs questionnaires. A Likert scale is the sum of responses on several Likert items. A Likert item is simply a statement that the respondent is asked to evaluate by giving it a quantitative value on any kind of subjective or objective dimension, with the level of agreement/disagreement being the dimension most commonly used.
  Study participants will be asked to rate their likelihood that they would want the same study medication again if they had second cataract surgery on an 11-point Likert scale of 0 (not likely at all) to 10 (extremely likely)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Martel Eye Medical Group, Rancho Cordova, California
  - Levenson Eye Associates, Jacksonville, Florida
  - Vance Thompson Vision, West Fargo, North Dakota

IPD SHARING:
Plan to Share IPD: No